CLINICAL TRIAL: NCT05240612
Title: A Clinical Pharmacological Study of MT-3921 in Subjects With Human T-cell Leukemia Virus Type 1 (HTLV-1)-Associated Myelopathy (HAM)
Brief Title: A Clinical Pharmacological Study of MT-3921 in Subjects With HTLV-1 Associated Myelopathy (HAM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-3921-C-101; jRCT2031210616 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2022-02-13; First posted 2022-02-15 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: HTLV-1-Associated Myelopathy (HAM)
MeSH Terms: conditions — Paraparesis, Tropical Spastic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MT-3921 (Experimental): Intravenous (IV)
  Interventions: Biological: MT-3921
- Placebo (Placebo Comparator): Intravenous (IV)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MT-3921 — Solution for infusion; Intravenous (IV)
  Other Names: Unasnemab
  Arms: MT-3921
Biological: Placebo — Solution for infusion; Intravenous (IV)
  Arms: Placebo

SUMMARY:
The purposes of this study is to assess the safety, tolerability, and pharmacokinetics of MT-3921 in subjects with Human T-cell Leukemia Virus Type 1 (HTLV-1)-Associated Myelopathy(HAM).

Subjects meeting eligibility criteria will enter the 6-month double-blind period. Subjects will be randomized in a 2:1 ratio to receive MT-3921 or placebo in a double blind manner.

ELIGIBILITY:
Inclusion Criteria:

Additional screening criteria check may apply for qualification:

* Subjects aged 20 years or older on the day of consent
* Subjects with a confirmed diagnosis of HAM according to the diagnostic algorithm of Practical Guideline for HAM 2019 on the day of consent
* Subjects with an Osame's motor disability score (OMDS) of ≥4 and ≤6 at Screening and on the first day of the Treatment period (predose)
* Subjects with no change in OMDS for at least 3 months before the day of consent
* Subjects with a CSF concentration neopterin of ≥6 pmol/mL at Screening
* Subjects on maintenance oral steroid therapy who have continued to receive the same dose equivalent to ≤10 mg/day of prednisolone for at least 3 months before the day of consent

Exclusion Criteria:

Additional screening criteria check may apply for qualification:

* Subjects who have a history of anaphylaxis or clinically significant allergic reactions due to administration of antibody products
* Subjects exhibiting or with a history of malignant tumor.
* Subjects with adult T-cell leukemia/lymphoma (ATL) or those with positive HTLV-1 clonality test (Southern blot) at screening and suspected of having ATL
* Subjects with spinal cord compression lesions, such as cervical spine disease, disc herniation, and ossification of the yellow ligament
* Subjects with psychiatric disorders, epileptic seizures, or dementia.
* Subjects with suicide attempts or suicidal ideation corresponding to item 4 or 5 on the Columbia Suicide Rating Scale (C-SSRS) at screening and/or on the first day of the Treatment period (predose)
* Subjects exhibiting or with a history of hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infection.
* Subjects with the novel Coronavirus disease 2019 (COVID-19)
* Subjects with severe illness
* Male or female subjects of childbearing potential who do not agree to use a contraceptive measure from the day of consent to 16 weeks after the last dose of the investigational medical product
* Female subjects who are pregnant, lactating, or may be pregnant
* Subjects who have received anti-repulsive guidance molecule (RGM) a antibody containing this investigational medical product
* Subjects who participated in other clinical studies (including clinical trials) and received drugs (including investigational medical products) or therapy within 12 weeks before the day of consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with adverse events | 36 weeks
Percentage of subjects with adverse reactions | 36 weeks
Serum concentrations of MT-3921 | PK samples will be collected at predose, 1.5 hours, 2, 4, 8, 12, 20 (predose and 1.5 hours), 24, 36 weeks post-dose.
CSF concentrations of MT-3921 | PK samples will be collected at 2, 4, 12, 24 weeks post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- St. Marianna University Hospital, Kawasaki-shi, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: No